CLINICAL TRIAL: NCT02207036
Title: Social Media Intervention for Young Adult Smokers
Brief Title: Tobacco Status Project: Social Media Intervention for Young Adult Smokers
Acronym: TSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A119678; 5K23DA032578 (NIH)
Record Dates: First submitted 2014-05-13; First posted 2014-08-01 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Smoking
Keywords: Tobacco; cigarettes; cessation; intervention; young adults; Internet; social media; mobile health
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Facebook intervention (Experimental): Assignment to private group on Facebook with 3 months of content delivered to the group.
  Interventions: Behavioral: Facebook intervention
- Referral (Active Comparator): Referral to smokefree.gov website
  Interventions: Behavioral: Smokefree.gov

INTERVENTIONS:
Behavioral: Facebook intervention — 90 days of Facebook messaging, weekly Ask the Doctor sessions
  Arms: Facebook intervention
Behavioral: Smokefree.gov — referral to the NCI Smokefree.gov website
  Arms: Referral

SUMMARY:
This randomized clinical trial will test the efficacy of a Facebook intervention based on the Transtheoretical Model (Prochaska and DiClemente) and US Public Health Service Clinical Practice Guidelines with young adults who smoke cigarettes who are age 18 to 25 (N=480).

DETAILED DESCRIPTION:
Participants will be randomized to one of two conditions: (1) a Facebook-delivered intervention tailored to readiness to quit smoking; or (2) the control condition (referral to the Smokefree.gov website). The intervention will include 12 weeks of Facebook-based messages and activities tailored to participants' stage of change.

Assessments will occur at baseline, 3, 6, and 12 months follow-up. Assessments will include measures on smoking patterns and thoughts about abstinence. All participants who report no past 7-day smoking will be asked to give biochemical verification of smoking status with saliva cotinine test kits that will be mailed to participants.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-25 years old
* english literate
* have access to Smartphone or computer with camera
* indicate they go on Facebook "most" (≥ 4) days per week
* have smoked ≥100 cigarettes in their lives and currently smoke at least 1 cigarette per day on 3 or more days of the week

Exclusion Criteria:

* do not read English
* younger than 18 or older than 25 years of age
* do not have access to a Smartphone or computer with a camera
* only go on Facebook 3 or fewer days a week
* have smoked less than 100 cigarettes in their lifetime or do not currently smoke at least 1 cigarette per day on 3 or more days of the week

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 501 (Actual)
Dates: Start 2014-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
7-day point prevalence abstinence at 3 months | 3 months post baseline
  Reports of no smoking in the 7 days prior to the 3 month assessment. Biochemical verification of abstinence will also be recorded.
7-day point prevalence abstinence at 6 months | 6 months post baseline
  Reports of no smoking in the 7 days prior to the 6 month assessment. Biochemical verification of abstinence will also be recorded.
7-day point prevalence abstinence at 12 months | 12 months post baseline
  Reports of no smoking in the 7 days prior to the 12 month assessment. Biochemical verification of abstinence will also be recorded.

SECONDARY OUTCOMES:
Reduction in cigarettes smoked by at least 50% between Baseline and each follow-up timepoint | 3, 6, and 12 months post baseline
  Reduction will be assessed at 3, 6, and 12 month follow-ups.
Quit attempts | 3, 6, and 12 month post-baseline
  Quit attempt during the follow-up period at 3, 6, and 12 months post-baseline.

OTHER OUTCOMES:
Health risk behaviors | 3, 6, and 12 months post baseline
  We will assess prevalence rates of health risk behaviors other than smoking including recent alcohol and illicit drug use, poor sleep quality, sedentary behavior, poor diet, depression, and high risk sexual behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle A Ramo, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco Department of Psychiatry, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramo DE, Liu H, Prochaska JJ. A mixed-methods study of young adults' receptivity to using Facebook for smoking cessation: if you build it, will they come? Am J Health Promot. 2015 Mar-Apr;29(4):e126-35. doi: 10.4278/ajhp.130326-QUAL-128. Epub 2014 Feb 27. PMID 24575728
- [Background] Ramo DE, Thrul J, Delucchi KL, Ling PM, Hall SM, Prochaska JJ. The Tobacco Status Project (TSP): Study protocol for a randomized controlled trial of a Facebook smoking cessation intervention for young adults. BMC Public Health. 2015 Sep 15;15:897. doi: 10.1186/s12889-015-2217-0. PMID 26374203
- [Background] Ramo DE, Thrul J, Chavez K, Delucchi KL, Prochaska JJ. Feasibility and Quit Rates of the Tobacco Status Project: A Facebook Smoking Cessation Intervention for Young Adults. J Med Internet Res. 2015 Dec 31;17(12):e291. doi: 10.2196/jmir.5209. PMID 26721211
- [Result] Ramo DE, Rodriguez TM, Chavez K, Sommer MJ, Prochaska JJ. Facebook Recruitment of Young Adult Smokers for a Cessation Trial: Methods, Metrics, and Lessons Learned. Internet Interv. 2014 Apr;1(2):58-64. doi: 10.1016/j.invent.2014.05.001. PMID 25045624
- [Derived] Ramo DE, Thrul J, Vogel EA, Delucchi K, Prochaska JJ. Multiple Health Risk Behaviors in Young Adult Smokers: Stages of Change and Stability over Time. Ann Behav Med. 2020 Jan 24;54(2):75-86. doi: 10.1093/abm/kaz025. PMID 31157881
- [Derived] McKelvey K, Ramo D. Conversation Within a Facebook Smoking Cessation Intervention Trial For Young Adults (Tobacco Status Project): Qualitative Analysis. JMIR Form Res. 2018 Sep 4;2(2):e11138. doi: 10.2196/11138. PMID 30684432